CLINICAL TRIAL: NCT05815121
Title: Interest of Acupressing in the Treatment of Preoperative Anxiety and Comfort of Patients Undergoing Oocyte Retrieval in Outpatient Surgery
Brief Title: Use of Acupressing in Reproductive Medicine
Acronym: ambauric
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hopital Foch (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2021_0165
Record Dates: First submitted 2023-02-08; First posted 2023-04-18 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-04

CONDITIONS: Fertility Disorders; Anxiety State
Keywords: Acupressing; oocyte; women; fertility
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Randomized, parallel goup, single
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Acupressing group (Experimental): Patients benefit from one session of acupressing with placement of 4 vaccaria seeds covered with stickers on the ears and 2 on the wrists.
  They will also be asked to regularly and gently massage the treated points
  Interventions: Other: Acupressing
- SHAM group (Sham Comparator): Patients treated according to the same scheme as the experimental group, but with stickers only on the points, and the points should not be massaged.
  Interventions: Other: Control

INTERVENTIONS:
Other: Acupressing — Acupuncture with placement of 4 vaccaria seeds covered with stickers on the ears and 2 on the wrists.
  Arms: Acupressing group
Other: Control — with stickers only on the points, and the points should not be massaged.
  Arms: SHAM group

SUMMARY:
The objective of this preliminary study is therefore to assess the feasibility, safety and reduction of perioperative anxiety thanks to acupressing. In addition, patients undergoing oocyte retrieval often present postoperatively with nausea, abdominal pain and discomfort. Acupuncture could also help these patients.

DETAILED DESCRIPTION:
Infertility can lead to the realization of follicular puncture or oocytes in order to obtain an embryo for medically assisted procreation. It is a long treatment for the couples concerned and this intervention, relatively simple in young patients, is associated with a very high level of anxiety. According to studies, the incidence of preoperative anxiety ranges from 11% to 80% in adult patients. In patients undergoing outpatient surgery, anxiolytics are not administered before anesthesia in outpatient surgery, as this would risk altering their "fitness for the street" and preventing their return home. Studies have shown a benefit of acupressing in the treatment of preoperative anxiety. This technique could therefore be an alternative to drug anxiety before surgery. Acupressing could also help these patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years old
* Scheduled to undergo an oocyte retrieval in outpatient surgery
* Anxiety score ≥ 3 when they arrived in the outpatient unit
* Subject is willing and able to provide informed consent
* Covered by a national healthcare insurance

Non-Inclusion Criteria:

* Ear's pavilion infection
* Wrist infection
* Previous treatment with auriculotherapy or acupuncture
* With a planned intervention that does not allow the delay of 45 min delay (+/- 15 min) between the acupuncture treatment and the STAI assessment
* Being deprived of liberty or under guardianship

Exclusion criteria

* Patient having recourse to any treatment or method of anxiolysis the morning of the procedure, after having given her consent
* Patient wishing to withdraw from the study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Femal with 18 years and older
Enrollment: 82 (Actual)
Dates: Start 2023-02-09 (Actual); Primary Completion 2023-03-11 (Actual); Study Completion 2023-03-11 (Actual)

PRIMARY OUTCOMES:
Anxiety assessement using State-Trait Anxiety Inventory questionnaire between baseline and 45 minutes after treatment. | Baseline to 45 minutes after treatment
  Anxiety assessed by the State-Trait Anxiety Inventory questionnaire. It consists of an auto-administered test of 20 items evaluating each item from 0 to 3 on the Likert scale (0= almost never, 1 = sometimes, 2 = often, 3 = almost always).
  The primary endpoint is the absolute difference in the state anxiety score measured between the baseline measurement and the measurement 45 minutes after treatment.

SECONDARY OUTCOMES:
Absolute difference measurement between the baseline and the immediate preoperative measurement | between baseline to the immediate preoperative measurement
  Anxiety score measured by numeric scale (0-10). 0 corresponding to no anxiety and 10 more anxiety
Absolute difference measurement between inclusion and when leaving the recovery room | before procedure to time when leaving the recovery room (up to 2 hours)
  Anxiety score measured by numeric scale (0-10). 0 corresponding to no anxiety and 10 more anxiety
Absolute difference measurement between baseline and day 1 | up 24 hours after treatment
  Anxiety score measured by numeric scale (0-10). 0 corresponding to no anxiety and 10 more anxiety
Pain score measured by numeric scale when leaving the recovery room | When leaving the recovery room (up to 2 hours)
  Pain score measured by numeric scale (0-10). 0 corresponding to no pain and 10 more pain
Postoperative nausea and vomiting occurring | In the recovery room (up to 2 hours)
  Proportion of patients declaring postoperative nausea and vomiting occurring during the stay in the recovery room
Postoperative retention of urine | In the recovery room (up to 2 hours)
  Proportion of patients declaring retention of urine or the need for catheterization for absence or delay in urination occurring during the stay in the recovery room
Tolerance of acupressing treatment | In the recovery room (up to 2 hours)
  The presence or absence of pain and discomfort in the recovery room attributed to the treatment of acupuncture by the patient
Satisfaction questionnaire | In the recovery room (up to 2 hours)
  Proportion of patients answering yes to the question "if you had to do it again, would you choose the same technique?" " when leaving the recovery room
Quality of sleep measurement | up 24 hours after treatment
  Quality of sleep measured using the SPIEGEL questionnaire the day after treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Mireille MICHEL-CHERQUI, MD, Principal Investigator — Foch Hospital; Sabrina MA HAR, MD, Study Director — Foch Hospital
Locations (1):
- Foch Hospital, Suresnes, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Villa G, Lanini I, Amass T, Bocciero V, Scire Calabrisotto C, Chelazzi C, Romagnoli S, De Gaudio AR, Lauro Grotto R. Effects of psychological interventions on anxiety and pain in patients undergoing major elective abdominal surgery: a systematic review. Perioper Med (Lond). 2020 Dec 8;9(1):38. doi: 10.1186/s13741-020-00169-x. PMID 33292558
- [Background] Williams JB, Alexander KP, Morin JF, Langlois Y, Noiseux N, Perrault LP, Smolderen K, Arnold SV, Eisenberg MJ, Pilote L, Monette J, Bergman H, Smith PK, Afilalo J. Preoperative anxiety as a predictor of mortality and major morbidity in patients aged >70 years undergoing cardiac surgery. Am J Cardiol. 2013 Jan 1;111(1):137-42. doi: 10.1016/j.amjcard.2012.08.060. PMID 23245838
- [Background] Oleson TD, Kroening RJ, Bresler DE. An experimental evaluation of auricular diagnosis: the somatotopic mapping or musculoskeletal pain at ear acupuncture points. Pain. 1980 Apr;8(2):217-229. doi: 10.1016/0304-3959(88)90009-7. PMID 7402685
- [Background] Usichenko TI, Hua K, Cummings M, Nowak A, Hahnenkamp K, Brinkhaus B, Dietzel J. Auricular stimulation for preoperative anxiety - A systematic review and meta-analysis of randomized controlled clinical trials. J Clin Anesth. 2022 Feb;76:110581. doi: 10.1016/j.jclinane.2021.110581. Epub 2021 Nov 12. PMID 34781116
- [Background] Saku K, Mukaino Y, Ying H, Arakawa K. Characteristics of reactive electropermeable points on the auricles of coronary heart disease patients. Clin Cardiol. 1993 May;16(5):415-9. doi: 10.1002/clc.4960160509. PMID 8504576
- [Background] Ceccherelli F, Gagliardi G, Seda R, Corradin M, Giron G. Different analgesic effects of manual and electrical acupuncture stimulation of real and sham auricular points: a blind controlled study with rats. Acupunct Electrother Res. 1999;24(3-4):169-79. doi: 10.3727/036012999816356309. PMID 10768414
- [Background] He W, Wang X, Shi H, Shang H, Li L, Jing X, Zhu B. Auricular acupuncture and vagal regulation. Evid Based Complement Alternat Med. 2012;2012:786839. doi: 10.1155/2012/786839. Epub 2012 Nov 27. PMID 23304215
- [Background] Usichenko TI, Mustea A, Pavlovic D. On ears and Head. Acupunct Med. 2010 Dec;28(4):165-6. doi: 10.1136/aim.2010.003244. No abstract available. PMID 21148074
- [Background] Mora B, Iannuzzi M, Lang T, Steinlechner B, Barker R, Dobrovits M, Wimmer C, Kober A. Auricular acupressure as a treatment for anxiety before extracorporeal shock wave lithotripsy in the elderly. J Urol. 2007 Jul;178(1):160-4; discussion 164. doi: 10.1016/j.juro.2007.03.019. Epub 2007 May 17. PMID 17499304
- [Background] Qu F, Zhang D, Chen LT, Wang FF, Pan JX, Zhu YM, Ma CM, Huang YT, Ye XQ, Sun SJ, Zheng WJ, Zhang RJ, Xu J, Xing LF, Huang HF. Auricular acupressure reduces anxiety levels and improves outcomes of in vitro fertilization: a prospective, randomized and controlled study. Sci Rep. 2014 May 22;4:5028. doi: 10.1038/srep05028. PMID 24848522
- [Background] Williams VS, Morlock RJ, Feltner D. Psychometric evaluation of a visual analog scale for the assessment of anxiety. Health Qual Life Outcomes. 2010 Jun 8;8:57. doi: 10.1186/1477-7525-8-57. PMID 20529361
- [Background] Tian M, Huang Y, Wang X, Cao M, Zhao Z, Chen T, Yuan C, Wang N, Zhang B, Li C, Zhou X. Vaccaria segetalis: A Review of Ethnomedicinal, Phytochemical, Pharmacological, and Toxicological Findings. Front Chem. 2021 Apr 29;9:666280. doi: 10.3389/fchem.2021.666280. eCollection 2021. PMID 33996757
- [Background] Nielsen A, Gereau S, Tick H. Risks and Safety of Extended Auricular Therapy: A Review of Reviews and Case Reports of Adverse Events. Pain Med. 2020 Jun 1;21(6):1276-1293. doi: 10.1093/pm/pnz379. PMID 32430505
- [Background] Wang SM, Maranets I, Weinberg ME, Caldwell-Andrews AA, Kain ZN. Parental auricular acupuncture as an adjunct for parental presence during induction of anesthesia. Anesthesiology. 2004 Jun;100(6):1399-404. doi: 10.1097/00000542-200406000-00011. PMID 15166558